CLINICAL TRIAL: NCT01330563
Title: Drug-Drug Interaction Study to Investigate the Effect of Ketoconazole on the Pharmacokinetic Properties of CKD-501 in Healthy Male Volunteer: Open, Randomised, 2-way Crossover, Clinical Trial
Brief Title: Drug-drug Interaction Study (CKD-501, Ketoconazole)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Chong Kun Dang Pharmaceutical, Chin Kim
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19HPS11G
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug-Drug interaction between the CKD-501 and ketoconazole
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-501 (Experimental): Subjects received Ketoconazole 200 mg twice daily for 5 days in one period and in the other period, Subjects don't receive Ketoconazole.
  In addition, The CKD-501 is administered on day 5
  Interventions: Drug: CKD-501, Ketoconazole
- ketoconazole (Experimental): Subjects received Ketoconazole 200 mg twice daily for 5 days in one period and in the other period, Subjects don't receive Ketoconazole.
  In addition, The CKD-501 is administered on day 5
  Interventions: Drug: CKD-501, Ketoconazole

INTERVENTIONS:
Drug: CKD-501, Ketoconazole — Subjects received single 0.5mg doses of CKD-501 alone in one period and, in the other period, Ketoconazole 200 mg twice daily for 5 day with the CKD-501 dose also co-administered with Ketoconazole on day 5.
  Other Names: Lobeglitazone, Ketoconazole

SUMMARY:
The purpose of this study is to assess the effect of Ketoconazole on the pharmacokinetic characteristics of CKD-501 in healthy subject.

DETAILED DESCRIPTION:
From day 1 to day 5, Ketoconazole 200mg is administered twice daily to Group 1 patients during period 1. Then on day 5,CKD-501 0.5mg is co-administered Group 1 patients at period 1. After 28 day-break, period 2 will CKD-501 0.5mg administered on day 5. Period 2 will not Ketoconazole administered.

Group 2 is administered in reverse order.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 aged and 45 years old in healthy males
* 18.5 ≤ IBW < 25
* Agreement with written informed consent

Exclusion Criteria:

* Hypersensitivity reactions to drugs or clinically significant hypersensitivity reactions in the history of party
* Medication with drug-mediated induction/inhibition metabolic enzyme such as Midazolam within 1 month or with may affect the clinical trial
* Subject has taken abnormal meals which affects the ADME of drug
* Subject has a history(such as gastric or duodenal ulcer, gastrointestinal surgical histories except for an appendectomy) affects the ADME of drug
* Substance abuse, or a history of drug abuse showed a positive for the party
* Continued to be taking caffeine (caffeine > 5 cup/day), drinking (alcohol > 210 g/week) or cannot stop drinking or severe heavy smoker(cigarette > 10 cigarettes per day)during clinical trials
* Previously participated in other trial within 60 days
* Previously donate whole blood within 60 days or component blood within 30 days
* Inadequate subject by medical examination(medical history, physical examination, ECG, laboratory test) within 28 days of starting administration of investigational drug
* SBP >140 mmHg, SBP < 90 mmHg or DBP > 90 mmHg, DBP < 50 mmHg or Pulse > 100 per/min, Pulse < 50 per/min
* 12-lead ECG, QTc > 450 msec
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
CKD-501 AUC | 0(Day 5), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48hr

SECONDARY OUTCOMES:
CKD-501 Cmax | 0(Day 5), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48hr
CKD-501 Tmax | 0(Day 5), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48hr

CONTACTS AND LOCATIONS:
Overall Officials: Minsoo Park, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Sil Oh E, Ok Kim C, Kim KH, Kim YN, Kim C, Lee JI, Park MS. Effect of ketoconazole on lobeglitazone pharmacokinetics in Korean volunteers. Clin Ther. 2014 Jul 1;36(7):1064-71. doi: 10.1016/j.clinthera.2014.05.064. PMID 25047497